CLINICAL TRIAL: NCT05921578
Title: Cone-beam CT in the Diagnosis and Surgical Treatment of Otosclerosis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Steven Andersen, M.D., PhD, Senior Researcher, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-22067452
Record Dates: First submitted 2023-06-06; First posted 2023-06-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Otosclerosis; Cone Beam Computed Tomography; Stapes Fixation
Keywords: otosclerosis; stapedotomy; cone beam CT
MeSH Terms: conditions — Otosclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine diagnostic workup (No Intervention)
- Routine diagnostic workup + pre-operative CBCT-based planning (Experimental)
  Interventions: Diagnostic Test: Pre-operative planning based on CBCT

INTERVENTIONS:
Diagnostic Test: Pre-operative planning based on CBCT — Pre-operative planning based on CBCT
  Arms: Routine diagnostic workup + pre-operative CBCT-based planning

SUMMARY:
Our studies will systematically investigate and establish evidence on whether Cone-beam computed tomography (CBCT) of the temporal bone could be used in the diagnosis and treatment of otosclerosis and in the post-operative follow-up after stapedotomy.

DETAILED DESCRIPTION:
Cone-beam CT has a high resolution and a low effective radiation dose to the patient when compared to conventional CT-scans. Surgical treatment of otosclerosis is primarily by stapedotomy. The decision of surgical treatment is currently based on the history, clinical examination, and audiological tests, but stapes fixation can only be confirmed per-operatively.

This protocol includes the following overall aims for the following studies:

* To establish the diagnostic precision of clinical CBCT in diagnosing otoslcerosis, i.e., the sensibility and specificity for our scanning protocols (n=50).
* To determine if CBCT can support the clinicians' decision making in the diagnosis of otosclerosis (n=100).
* To assess the value of CBCT in the planning of stapes surgery. Two groups will be established: CBCT-based pre-operative planning (e.g., prothesis parameters and anatomic landmarks) and no-planning (standard treatment). Patients will be allocated by 1:1 randomization (n=75).
* To assess the value of CBCT in the post-operative follow-up of 2-3 weeks, 2-3 months, and 12 months. Follow-up includes a clinical examination, audiometry, CBCT (block-randomized), and patient questionnaires (audiometry and patient questionnaire not at the "2-3 weeks" control) (n=75).
* To assess the value of pre-preoperative CBCT on post-surgical result at follow up (2-3 weeks, 2-3, months and 12-months) (n=75).

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years of age).
* Referred to our department suspected for otosclerosis.
* Consents to participation in the project.

Exclusion Criteria:

* A history of surgical treatment for otosclerosis (ipsilateral ear).
* A history of tympanoplasty type 2-4 (ipsilateral ear).
* Other competing middle-ear diseases (ipsilateral ear).

Inclusion and exclusion criteria for patients enrolled for post-surgical follow-up are the same as above in addition to:

Exclusion:

- Intraoperative findings not supporting otosclerosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic precision of CBCT of the temporal bone in diagnosing otosclerosis. | Per-operative
  The diagnostic precision will be established, i.e., the sensibility and specificity for our scanning protocols.
Clinical decision-making in the diagnosis of suspected otosclerosis | Baseline
  The proportion of patients where CBCT assists in the decision clinical decision making of otosclerosis.
Prothesis placement (pre-operative planning) | 12 months
  Pre-operative CBCT based planning on the prothesis placement at surgery.
Post-operative follow-up: patient reported hearing | 12 months
  The effect of pre-operative planning on the patient reported hearing at follow-up.
Post-operative follow-up: measured hearing | 12 months
  The effect of pre-operative planning on the measured hearing (audiometry) at follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No